CLINICAL TRIAL: NCT01811225
Title: Smoking, Sex Hormones, and Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2012NTLS018
Record Dates: First submitted 2013-02-21; First posted 2013-03-14 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Nicotine Dependence; Contraception
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-Dose Contraceptive, then High-Dose (Experimental): Females, 18-35 years old, non-pregnant, using oral contraceptive for at least the last 3 months before enrollment will be given Tri-Sprintec and generic Prometrium.
  Participants in this arm will begin with the "low" dose progesterone, which is seven days of placebo Tri-sprintec + placebo generic Prometrium twice daily (7AM and 7PM). Then participants in this arm will move to the "high" dose progesterone, which is seven days of placebo Tri-Sprintec + 200mg of generic Prometrium twice daily (7AM and 7PM).
  Interventions: Drug: Low-dose Progesterone; Drug: High-dose Progesterone
- High-Dose Contraceptive, then Low-Dose (Experimental): Females, 18-35 years old, non-pregnant, using oral contraceptive for at least the last 3 months before enrollment will be given Tri-Sprintec and generic Prometrium.
  Participants in this arm will begin with the "high" progesterone dose, which is seven days of placebo Tri-Sprintec + 200mg of generic Prometrium twice daily (7AM and 7PM). Then participants in this arm will move to the "low" dose progesterone, which is seven days of placebo Tri-sprintec + placebo generic Prometrium twice daily (7AM and 7PM).
  Interventions: Drug: Low-dose Progesterone; Drug: High-dose Progesterone

INTERVENTIONS:
Drug: Low-dose Progesterone — The "low" progesterone dose is seven days of placebo Tri-sprintec + placebo generic Prometrium twice a day (7AM and 7PM).
Drug: High-dose Progesterone — The "high" progesterone dose is seven days of placebo Tri-Sprintec + 200mg of generic Prometrium twice a day (7AM and 7PM).

SUMMARY:
The investigators aim to (1) examine the association between levels of progesterone (Prog), allopregnanolone (Allo), and the estradiol/progesterone (E2/P) ratios with smoking-related symptomatology during ad libitum smoking and (2) determine the association between Prog, Allo, and E2/P with the changes in smoking-related symptomatology and response to nicotine following overnight abstinence

DETAILED DESCRIPTION:
The sample population will consist of oral contraceptive users, both "low" and "high" dose levels of exogenous progesterone with a consistent dose of exogenous estrogen. Participants will complete data collection procedures including providing saliva (cortisol to measure stress), urine (cotinine and 3-Hydroxycotinine to measure nicotine exposure), and blood (progesterone, allopregnanolone, and estradiol) samples, as well as ecological momentary assessments (EMA) daily for seven-days. Participants will also complete a 3-hour smoking topography lab session after overnight abstinence and a 4.5-hour nicotine nasal spray lab session after a 14-hour abstinence. These sessions will contain a nicotine challenge via smoking a cigarette or nasal spray with timed-series physiological, subjective, and behavioral responses.

ELIGIBILITY:
Inclusion Criteria:

* currently taking oral contraceptives
* English fluency
* Ability to provide informed consent

Exclusion Criteria:

* use of progestin only contraceptive
* pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2012-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S. Allen, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Allen S, Harrison K, Petersen A, Goodson J. Smoking-related symptomatology in pregnant smokers during ad libitum smoking and following overnight smoking abstinence. BMC Res Notes. 2019 Aug 1;12(1):473. doi: 10.1186/s13104-019-4503-x. PMID 31370907

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Low-Dose Contraceptive, Then High-Dose | High-Dose Contraceptive, Then Low-Dose
Started | 49 | 46
Completed | 24 (53 completed one arm of the cross-over and 43 completed two arms of the cross-over) | 29
Not Completed | 25 | 17
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 12 | 8
Not completed — transporation | 1 | 0
Not completed — unable to remain smoke free overnight | 10 | 6
Period: Treatment Period 2
Arm/Group | Low-Dose Contraceptive, Then High-Dose | High-Dose Contraceptive, Then Low-Dose
Started | 24 | 29
Completed | 20 | 23
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — unable to remain smoke free overnight | 3 | 4

BASELINE CHARACTERISTICS:
Population: This is cross-over study. Baseline data is presented as a pool of all participants at baseline.
Groups:
- All Participants: All participants at baseline
Arm/Group | All Participants
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 12
  White | 41
  Native American | 5
  Asian | 2
  Mixed Race | 9
  Hawaiian/Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Smoking Urges
Description: Questionnaire on Smoking Urges-Brief (QSU-Brief): This ten-item version of the original form (QSU) was developed by Tiffany and Drobes and has an excellent level of reliability (α = .97). Total QSU-Brief. Scores can average between 1-7. A higher scores means more urges.
Time Frame: after overnight abstinence on day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low-Dose Contraceptive: Females, 18-35 years old, non-pregnant, using oral contraceptive for at least the last 3 months before enrollment will be given a low-dose contraceptive.
  The "low" progesterone dose is seven days of placebo Tri-sprintec + placebo generic Prometrium twice a day (7AM and 7PM).
- High-Dose Contraceptive: Females, 18-35 years old, non-pregnant, using oral contraceptive for at least the last 3 months before enrollment will be given a high-dose contraceptive.
  The "high" progesterone dose is seven days of placebo Tri-Sprintec + 200mg of generic Prometrium twice a day (7AM and 7PM).
Arm/Group | Low-Dose Contraceptive | High-Dose Contraceptive
Number analyzed (Participants) | 34 | 36
score on a scale | 5.0 (1.4) | 5.5 (2.1)

2. Secondary Outcome: Change in Positive and Negative Affect Scale Following Overnight Abstinence
Description: Positive and Negative Affect Scale (PANAS): Participants rate 20 words associated with positive or negative affect using a five-point Likert-type scale. This scale has been shown to have high internal consistency. Positive PANAS scores can range from 10-50. A higher score means greater positive affect. Negative PANAS score can range from 10-50. A higher score means greater negative affect.
Time Frame: after overnight abstinence on day 8
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low-Dose Contraceptive | High-Dose Contraceptive
Number analyzed (Participants) | 34 | 36
score on a scale
  Positive Affect | 26.21 [10 to 50] | 24.09 [10 to 50]
  Negative Affect | 17.01 [10 to 42] | 15.41 [10 to 37]

3. Secondary Outcome: Change in Cohen Perceived Stress Scale
Description: Cohen Perceived Stress Scale (PSS): This ten-item questionnaire has been validated in a variety of populations including pregnant and postpartum women. It uses five-items to assess ten questions resulting in two factors negative feelings and inability to handle stress. It has high internal reliability (alpha = 0.75). Score range from 0-56. A higher score means more perceived stress.
Time Frame: after overnight abstinence on day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Dose Contraceptive | High-Dose Contraceptive
Number analyzed (Participants) | 34 | 36
score on a scale | 14 (4.3) | 15 (3.8)

ADVERSE EVENTS:
Time Frame: AE were collected from oral contraceptive users over 3 months
Arm/Group | Low-Dose Contraceptive | High-Dose Contraceptive
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 19/34 | 17/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Contraceptive (N=34) | High-Dose Contraceptive (N=36)
pain (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Vomiting (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Cold and Sinus infection (Infections and infestations) | 3 (3) | 1 (1)
Breast Tenderness or soreness (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2)
Dizzy lightheaded (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 7 (7) | 5 (5)
Restless legs (General disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT01811225/Prot_SAP_000.pdf